CLINICAL TRIAL: NCT04448912
Title: Damage-Control Surgery in Patients With Non-traumatic Abdominal Emergencies: A Systematic Review and Meta-Analysis
Brief Title: Meta-Analysis on Damage Control Surgery in Patients With Non-Traumatic Abdominal Emergencies
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: SRMA non-trauma DCS
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Damage Control Surgery; Non-traumatic Abdominal Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-trauma damge control surgery: Patients with non-traumatic abdominal emergencies undergoing damage control surgery.
  Interventions: Procedure: Damage control surgery
- Non-trauma conventional surgery: Patients with non-traumatic abdominal emergencies undergoing conventional surgery with primary abdominal closure.
  Interventions: Procedure: Conventional surgery

INTERVENTIONS:
Procedure: Damage control surgery — Surgery for non-traumatic abdominal emergencies using the damage control approach
  Groups: Non-trauma damge control surgery
Procedure: Conventional surgery — Conventional surgery for non-traumatic abdominal emergencies
  Groups: Non-trauma conventional surgery

SUMMARY:
This systematic review and meta-analysis aims to investigate the effect of damage-control surgery on mortality in patients with non-traumatic abdominal emergencies. Literature search will be conducted using PubMed. Two meta-analyses will be performed comparing (1) mortality in patients with non-trauma damage control surgery vs. non-trauma conventional surgery and (2) the observed vs. expected mortality rate in patients undergoing non-trauma damage-control surgery.

DETAILED DESCRIPTION:
After the successful implementation in trauma patients, damage control surgery (DCS) is being increasingly used in patients with non-traumatic abdominal emergencies, too. However, non-trauma DCS is an ongoing matter of debate as the open abdomen treatment typically performed in DCS is a non-anatomical situation and associated with potentially severe side effects. To date, DCS in patients with non-traumatic abdominal emergencies has not yet been comprehensively assessed in meta-analysis.

A systematic literature search will be conducted using the National Library of Medicine's Medline database (PubMed). The search strategy will be based on the PICOS process. Original research articles in English language addressing (1) mortality in patients undergoing non-trauma DCS vs. non-trauma conventional surgery or (2) the observed vs. expected mortality in non-trauma DCS will be included.

Two meta-analyses will be performed, comparing (1) mortality in patients undergoing non-trauma DCS vs. non-trauma conventional surgery and (2) the observed vs. expected mortality rate in patients undergoing non-trauma DCS based on outcome prediction scores. Meta-analysis will be performed using a random-effects model. The estimated effect size for mortality will be reported as risk difference with 95% confidence intervals. Sensitivity analysis will be performed by repeating the analysis in the subgroups of studies with the same study design and studies that applied the same outcome prediction score.

ELIGIBILITY:
Inclusion Criteria:

* Articles on damage control surgery in patients with non-traumatic abdominal emergencies
* Reported in-hospital or 30-day mortality in patients undergoing non-trauma damage control surgery vs non-trauma conventional surgery or
* Reported observed in-hospital or 30-day mortality vs expected mortality in patients undergoing non-trauma damage control surgery
* Articles published from 2000 to 2020
* Articles including patients older than 18 years
* Original research articles
* Articles in English language

Exclusion Criteria:

* Articles describing trauma patients exclusively
* Articles describing pediatric patients (age below or equal to 18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for non-traumatic abdominal emergencies.
Sampling Method: Non-Probability Sample
Enrollment: 2170 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-04-24 (Actual)

PRIMARY OUTCOMES:
Mortality | From hospital admission to discharge, expected to be up to 4 weeks
  Death after surgery for non-traumatic abdominal emergencies

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Haltmeier, MD, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern University Hospial, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haltmeier T, Falke M, Quaile O, Candinas D, Schnuriger B. Damage-control surgery in patients with nontraumatic abdominal emergencies: A systematic review and meta-analysis. J Trauma Acute Care Surg. 2022 Jun 1;92(6):1075-1085. doi: 10.1097/TA.0000000000003488. Epub 2021 Dec 9. PMID 34882591